CLINICAL TRIAL: NCT05192499
Title: Respiratory Dysbiosis in Preschool Children with Asthma: Predictive of a Severe Form
Acronym: DREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC21.0252
Record Dates: First submitted 2021-11-16; First posted 2022-01-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Asthma in Children; Dysbiosis
Keywords: Paediatric Pulmonology; asthma; respiratory microbiome
MeSH Terms: conditions — Dysbiosis; Asthma | interventions — Occult Blood; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Exploratory multicentric prospective case-controlled study
Masking Description: DREAM is a case-controlled study in open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Other): Patients aged to 1 to 3 years with severe asthma (i.e. resistant to inhaled corticosteroid doses less than or equal to 200μg fluticasone equivalent).
  "Severe" asthma patients (cases) are defined by poor asthma control under doses of inhaled corticosteroids ≤200μg fluticasone equivalent.
  Interventions: Procedure: Stool test; Procedure: Blood test; Procedure: Induced sputum; Procedure: nasale virology
- Control (Other): Patients aged to 1 to 3 years with low or moderate asthma (controlled with mild to moderate doses of inhaled corticosteroids less than or equal to 200μg of fluticasone equivalent).
  "Mild to moderate" asthma patients (controls) are defined by disease control by first-line treatment in asthma, i.e. corticosteroids inhaled at mild to moderate doses of ≤200 micrograms/day of fluticasone equivalent.
  Interventions: Procedure: Stool test; Procedure: Blood test; Procedure: Induced sputum; Procedure: nasale virology

INTERVENTIONS:
Procedure: Stool test — At inclusion (day 0), stools will be collected with a kit for to remove to 5 mg for each patient.
Procedure: Blood test — Blood sample taken during inclusion (day 0) will be collected. There is between 19 and 26 mL for each patient.
Procedure: Induced sputum — At inclusion (day 0), bronchial aspiration after inhalation induction of 4 mL of 6% salt serum administered (after 200 μg of salbutamol via an inhalation chamber during a bronchial drainage session).
Procedure: nasale virology — At inclusion (Day 0), patients will be taken nasal swab for virology with swab adapted for nasal swab or with suction trap when blowing the child's nose (depending on center practice)and multiplex PCR.

SUMMARY:
The prevalence of asthma in preschool children is between 11 and12%. Inhaled corticosteroid therapy is the main therapy used, however this treatment seems insufficiently effective in some children.

Recent research in cystic fibrosis has made it possible to highlight pulmotypes corresponding to the different stages of pulmonary dysbiosis, and a predictive microbiological signature of an increased risk of early primocolonization to P. aeruginosa. These pulmotypes are the result of the so-called "enterotyping" analysis, a biostatistical method that makes it possible to stratify individuals according to the analysis of the microbiota. In the light of these data, it seems interesting to transcribe the concept of using a biomarker of the microbiota in the monitoring of a chronic lung disease such as asthma.

The hypothesis is that there is respiratory dysbiosis causing corticosteroid resistance to treatment in children under 3 years of age with severe asthma.

DETAILED DESCRIPTION:
The prevalence of asthma in preschool children is estimated to between 11 and 12%.

Inhaled corticosteroid therapy is the main therapy used, however this treatment seems insufficiently effective in some children.

Recent research in cystic fibrosis has made it possible to highlight pulmotypes corresponding to the different stages of pulmonary dysbiosis, and a predictive microbiological signature of an increased risk of early primocolonization to P. aeruginosa. These pulmotypes are the result of the so-called "enterotypeing" analysis, a biostatistical method that makes it possible to stratify individuals according to the analysis of the microbiota. In the light of these data, it seems interesting to transcribe the concept of using a biomarker of the microbiota in the monitoring of a chronic lung disease such as asthma.

The hypothesis is that there is respiratory dysbiosis causing corticosteroid resistance to treatment in children under 3 years of age with severe asthma.

The goal of this study is to research a difference between respiratory dysbiosis and severe asthma (i.e. resistant to doses of inhaled corticosteroids less than or equal to 200μg of fluticasone equivalent).

DREAM is a exploratory multicentric prospective case-control study.

The primary objective is to research a difference between respiratory dysbiosis and severe asthma (i.e. resistant to doses of inhaled corticosteroids less than or equal to 200μg of fluticasone equivalent) in children less than 36 months of age.

The secondary objectives are :

1. To compare the bacterial pulmotypes of children under 36 months of age with severe asthma with children with mild or moderate asthma.
2. To look for microbial biomarkers associated with corticosteroid resistance
3. To assess the association between digestive dysbiosis and severe asthma (i.e. resistant to inhaled corticosteroid doses less than or equal to 200μg fluticasone equivalent)
4. To look for an association between digestive dysbiosis and respiratory dysbiosis
5. To constitute a biocollection (sputum, stool, blood) of children with asthma for future analysis

30 patients are expected to be included in two arms : 15 uncontrolled asthmatic patients at moderate doses of inhaled corticosteroids and 15 asthmatic patients controlled at mild to moderate doses of inhaled corticosteroids.

Inclusion period : 12 months. Duration of patient's participation: 6 years Total study duration: 7 years

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 1 year and less than 3 years
* Diagnosis of asthma by a pediatrician
* Parental consent
* Affiliation to the social security system

Exclusion Criteria:

* Chronic pathologies: congenital heart disease, immune deficiency, cystic fibrosis, bronchopulmonary dysplasia, encephalopathy, primary ciliary dyskinesia, laryngomalacia, digestive pathology requiring digestive surgery
* Premature < 34 SA
* Recent antibiotic therapy (< 7 days)
* Treatment with oral corticosteroid therapy within the previous 10 days.
* Patient whose parent(s) is (are) minor(s)

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Number of species in the microbial Community | Day 0
  The main evaluation is the comparison of respiratory biodiversity assessed using quantitative indices such as alpha diversity. Alpha diversity calculates the richness (number of species or OTU) by samples and how these OTUs are distributed (equitability). Richness will be measured with the Chao1 and equity with the Simpson index. The Shannon index is a composite measurethat allows us to have both information together, richness and equity in the same index.
Index of microbial similarity of samples | Day 0
  The main evaluation is the comparison of respiratory biodiversity assessed using quantitative indices such beta diversity. Beta diversity analysis allows samples to be compared with each other. It calculates a matrix of distances between samples with the Bray Curtis/ Unifrac methods, weighted or not/ Jaccard by presence/absence. Next, the Principal Coordinate Analysis (PCoA ) will be used, multidimensional scaling to reduce this matrix to 2/3 dimensions. The samples from similar groups look alike with this analysis will be used.

SECONDARY OUTCOMES:
Enterotyping analysis | Day 0
  Characterization of bacterial pulmotypes by so-called "enterotyping" analysis in asthmatic children under 36 months of age. The enterotyping technique is a multifactorial technique that aims to group species / OTUs regularly found together. Enterotypes can characterize states of health or dysbiosis in the lung or intestines. OTU groups are used to classify individuals according to their lung / intestinal bacteria. The enterotypes / pulmotypes are considered already present in the literature and use PCA-type analyses to identify these groups of OTUs.
Relative abundance | Day 0
  Relative abundance (expressed as a percentage) of each of the identified bacteriological taxa
Indices of diversity | Day 0
  Types of indices of diversity of bacterial taxa identified in the digestive microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.